CLINICAL TRIAL: NCT04899869
Title: Faecal Microbiota Transplantation in Irritable Bowel Syndrome: a Randomised, Double-blind Cross-over Study Utilising Mixed Microbiota From Healthy Donors
Brief Title: Faecal Microbiota Transplantation in Irritable Bowel Syndrome
Acronym: MISCEAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomayer University Hospital (Other)
Collaborators: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Pavel Kohout, Pavel Kohout, Assoc. Prof., MD, PhD., Thomayer University Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: INT_TN_001
Record Dates: First submitted 2021-05-19; First posted 2021-05-25 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Irritable Bowel Syndrome With Diarrhea; Irritable Bowel Syndrome Mixed
Keywords: IBS - D, IBS - M
MeSH Terms: interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: Each study subject will undergo two pairs of faecal microbiota transplantation eight weeks apart (a total of four enemas for each patient). Our study design has several specific features: (a) Two consecutive transfers were designed to improve study microbiota engraftment. Before the first of every transfer pairs, the subjects will receive a reduced dose of oral polyethylene glycol for partial bowel preparation. (b) To help discern potential carry-over effects, a placebo-only group was included; this also enables us to assess long-term effects of the intervention. (c) The transferred microbiota is identical throughout the study, having been mixed beforehand, aliquoted and deep frozen. Its alpha diversity was artificially increased by mixing stools from several donors. (d) Placebo is made of the same mixture by careful autoclaving.
Who Masked: Participant, Care Provider, Investigator
Masking Description: double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (active microbiota first) (Other): Patients will first receive two enemas of active study microbiota mixture (deep-frozen stored stool microbiota mixed from eight donors in order to increase its diversity), then after eight weeks they will receive two enemas with placebo.
  Interventions: Other: Faecal microbiota transplantation with active study microbiota first
- Group B (inactive microbiota first) (Other): Patients will first receive placebo, then the active study microbiota mixture.
  Interventions: Other: Faecal microbiota transplantation with inactive autoclaved study microbiota first
- Group C (inactive microbiota only) (Other): Patients will receive similarly timed enemas with placebos only.
  Interventions: Other: Faecal microbiota transplantation with inactive autoclaved study microbiota only

INTERVENTIONS:
Other: Faecal microbiota transplantation with active study microbiota first — 2x enema with active study microbiota; after 8 wks 2x enema with inactive autoclaved study microbiota
  Arms: Group A (active microbiota first)
Other: Faecal microbiota transplantation with inactive autoclaved study microbiota first — 2x enema with inactive autoclaved study microbiota; after 8 wks 2x enema with active study microbiota
  Arms: Group B (inactive microbiota first)
Other: Faecal microbiota transplantation with inactive autoclaved study microbiota only — 2x enema with inactive autoclaved study microbiota; after 8 wks 2x enema with inactive autoclaved study microbiota
  Arms: Group C (inactive microbiota only)

SUMMARY:
Irritable bowel syndrome (IBS) is the most common functional bowel disorder, being present in approximately 10% of adult Europoid population. The etiology of IBS is elusive. Literature indicates that modification of patients´colonic microbiota might ameliorate the condition. Here we test an intervention by faecal microbiota transplantation of artificially inflated microbiome diversity, versus autoclaved placebo.

DETAILED DESCRIPTION:
Three-groups, double-blind, placebo-controlled, randomised, cross-over study in adult patients diagnosed with IBS (diarrhoeal or mixed form) according to Rome IV criteria. Each study subject will undergo two pairs of faecal microbiota transplantation (a total of four enemas for each patient), with the pairs of transfers being eight weeks apart. The active intervention substance is a mixed stool microbiota derived from healthy individuals, screened for infectious diseases according to European consensus conference on faecal microbiota transplantation guidelines, and who were preselected for high alpha diversity of their microbiome and distance in community ordination from IBS patients microbiota. Placebo is the same mixture, inactivated by autoclaving.

ELIGIBILITY:
Inclusion Criteria:

* Diarrhea Predominant Irritable Bowel Syndrome (IBS-D) or Irritable Bowel Syndrome with mixed bowel habits (IBS-M) according to the Rome IV criteria

Exclusion Criteria:

* The use of antibiotics within one month prior to faecal microbiota transplantation
* The use of probiotics within one month prior to faecal microbiota transplantation
* History of inflammatory bowel disease or gastrointestinal malignancy, systemic autoimmune diseases (ongoing or in history)
* Previous abdominal surgery (other than appendectomy or cholecystectomy or hernioplasty or cesarean section)
* HIV infection or other active infection
* Renal or hepatic disease (both defined by biochemistry workup)
* Diabetes mellitus, abnormal thyroid functions not controlled by thyroid medications
* Bipolar disorder or schizophrenia (ongoing or history thereof), moderately severe depression defined by Patient Health Questionnaire-9 (PHQ-9) score > 15
* Anxiety defined by a Generalised Anxiety Disorder 7 (GAD7) score > 10
* Current pregnancy and lactation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2021-06-17 (Actual); Primary Completion 2024-03-27 (Actual); Study Completion 2024-04-29 (Actual)

PRIMARY OUTCOMES:
Change in the IBS severity symptom score (IBS-SSS) | The difference between the score at four weeks after the intervention (study weeks 5 or 13, respectively) and the baseline score (week -1 in 'Active microbiota first' group or week 8 in 'Inactive microbiota first' group)
  Change in the IBS severity symptom score (IBS-SSS) in the active microbiota group relative to the placebo group.

SECONDARY OUTCOMES:
The acute change in the IBS severity symptom score (IBS-SSS) | study weeks 3 and 11, respectively
  IBS-SSS between baseline and two weeks after intervention
The long-term change in the IBS severity symptom score (IBS-SSS) | baseline and study week 32
  IBS-SSS between baseline (week -1) and week 32. The long term change will compare placebo group to merged active study microbiota groups.
Change in number of loose stools per day | baseline and study week 32
  Change in number of loose stools per day in the active microbiota group relative to the placebo group
Change in stool consistency | baseline and study week 32
  Change in stool consistency evaluated by Bristol stool scale (type 3 and 4 - normal; types 1,2,5,6 and 7 - abnormal) in the active microbiota group relative to the placebo group
Change in abdominal pain | baseline and study week 32
  Change in abdominal pain measured by Visual Analogue Scale (VAS) (0 - no pain, 10 - worst pain) in the active microbiota group relative to the placebo group
Change in frequency of bloating per week | baseline and study week 32
  Change in frequency of bloating per week (as there is no standardised measurement, it will be reported as number of episodes per time unit, where the possible answers could be: no bloating, bloating once a week, twice a week, three times a week, four times a week, five times a week, six times a week, bloating daily, bloating daily and sometimes at night, bloating more than half of days, bloating continuously) in the active microbiota group relative to the placebo group
Change in Body Mass Index | baseline and study week 32
  Change in Body Mass Index (BMI in kg/m^2) in the active microbiota group relative to the placebo group
Change in waist circumference | baseline and study week 32
  Change in waist circumference (in centimeters) in the active microbiota group relative to the placebo group
Change in body fat mass estimated by skinfold thickness measuring | baseline and study week 32
  Change in body fat mass estimated by measuring combined skinfold thickness at given locations (biceps, triceps, subscapular, suprailiac) in millimetres in the active microbiota group relative to the placebo group
Change in body fat mass measured by bioelectrical impedance analysis | baseline and study week 32
  Change in body fat mass in the active microbiota group relative to the placebo group measured by bioelectrical impedance analysis (in %)
Change in faecal microbiome's alpha (within-sample) diversity | baseline and study week 32
  Change in faecal microbiome's alpha (within-sample) diversity in the active microbiota group relative to the placebo group measured by Chao index of alpha diversity (higher value means higher alpha-diversity)
Change in faecal microbiome's beta (between samples) diversity | baseline and study week 32
  Change in faecal microbiome's beta (between samples) diversity in the active microbiota group relative to the placebo group assessed by the quantitative Bray-Curtis index (more distant means more different bacterial composition) ordinated by nonmetric multidimensional scaling (NMDS)
Change in the quantity of single-cell protist Blastocystis | baseline and study week 32
  Change in the quantity of single-cell protist Blastocystis in the active microbiota group relative to the placebo group assessed by a specific quantitative polymerase chain reaction assay measured in genomic equivalents per microlitre DNA (the higher concentration means more of Blastocystis)
The psychological and well-being effects of the therapy (IBS-QoL) | baseline and study week 32
  The psychological and well-being effects of the therapy scored by IBS-QoL questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Kohout, Principal Investigator — Thomayer University Hospital, Prague, Czech Republic
Locations (1):
- Thomayer University Hospital, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Yes
Only the researchers involved in the study have access to the final study dataset (IBS-SSS, frequency of urgent defecations, Bristol stool scale, abdominal pain and bloating), which will be shared in an anonymised form via the Zenodo repository.
Supporting Information: Study Protocol, ICF, CSR

REFERENCES:
- [Derived] Hurych J, Vejmelka J, Hlinakova L, Kramna L, Larionov V, Kulich M, Cinek O, Kohout P. Protocol for faecal microbiota transplantation in irritable bowel syndrome: the MISCEAT study - a randomised, double-blind cross-over study using mixed microbiota from healthy donors. BMJ Open. 2022 Jun 27;12(6):e056594. doi: 10.1136/bmjopen-2021-056594. PMID 35760542